CLINICAL TRIAL: NCT03173534
Title: WATCHMAN for Patients With Atrial Fibrillation Undergoing Transcatheter Aortic Valve Replacement
Brief Title: WATCH-TAVR, WATCHMAN for Patients With Atrial Fibrillation Undergoing Transcatheter Aortic Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: samir kapadia (Other)
Collaborators: Boston Scientific Corporation (Industry); The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, samir kapadia, Study Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WATCH-TAVR
Record Dates: First submitted 2017-05-23; First posted 2017-06-02 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Aortic Valve Stenosis
MeSH Terms: conditions — Atrial Fibrillation; Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 allocation ratio to the following treatment arms TAVR + Medical Therapy (n=175) or simultaneous TAVR + WATCHMAN (n=175)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TAVR + Medical Therapy (Active Comparator): n=172 will undergo Transcatheter Aortic Valve Replacement (TAVR) alone with medical management for atrial fibrillation
  Interventions: Device: TAVR
- TAVR + WATCHMAN (Experimental): n=177 will undergo simultaneous Transcatheter Aortic Valve Replacement (TAVR) with a WATCHMAN device.
  Interventions: Device: WATCHMAN; Device: TAVR

INTERVENTIONS:
Device: WATCHMAN — WATCHMAN Device is composed of a self-expanding nitinol structure with a porous membrane on the proximal face. The implant device is delivered to the Left Atrial Appendage by femoral venous access and transseptal puncture to enter the left atrium.
  Arms: TAVR + WATCHMAN
Device: TAVR — Transcatheter Aortic Valve Replacement

SUMMARY:
To evaluate the safety and effectiveness of the left atrial appendage occlusion with WATCHMAN Device in prevention of stroke and bleeding in patients with atrial fibrillation (AF) undergoing transcatheter aortic valve replacement (TAVR).

DETAILED DESCRIPTION:
WATCH-TAVR is a prospective, multicenter, randomized controlled trial. Only centers with approval for commercial WATCHMAN implantation will be included in this trial. Subjects will be enrolled at up to 32 centers in the United States. There will be up to 350 subjects enrolled, with 175 patients randomized to TAVR + medical therapy and 175 patients randomized to simultaneous TAVR+WATCHMAN to accumulate the necessary 191 primary events. Enrollment is expected to occur over the course of 18 months. Patients will be followed for a total of 2 years. Patients with non-valvular AF undergoing standard of care commercial TAVR will be enrolled in the trial.

For patients who receive the WATCHMAN device, plan of care will follow WATCHMAN labeling.Patients randomized to receive the WATCHMAN device will receive anticoagulation with warfarin and aspirin for 6 weeks after the procedure. After 6 weeks, the plan of care will follow WATCHMAN labeling. Patients randomized to the TAVR + medical therapy arm will be treated in accordance with standard of care with either warfarin, other anticoagulant/antiplatelet therapy, or no anticoagulation at the discretion of the treating physician. All patients will continue to receive routine post-TAVR follow-up and care.Patients will be monitored for primary and secondary endpoints as outlined. Baseline information and laboratory data will be collected as described in the protocol.

At trial conclusion, total number of subjects enrolled was 349. There were 172 subjects enrolled in the TAVR + Medical Therapy arm and 177 subjects enrolled in the TAVR + WATCHMAN arm.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age.
2. The patient meets criteria for and is scheduled to undergo TAVR procedure
3. The patient has documented paroxysmal, persistent, or permanent atrial fibrillation.
4. The patient meets the WATCHMAN labeling guidelines and is eligible to undergo the WATCHMAN implantation procedure.
5. The patient is eligible for short term warfarin therapy.
6. The patient or legal representative is able to understand and willing to provide written informed consent to participate in the trial.
7. The patient is able and willing to return for required follow-up visits and examinations.

Exclusion Criteria:

1. The patient had a stroke or TIA within the last 6 months prior to enrollment.
2. Contraindication for short term anticoagulation.

3 .Moderate or severe Mitral Stenosis with mean gradient across Mitral Valve >10 mm Hg or Mitral Valve Area < 1.2cm2.

4. The patient has symptomatic carotid disease (i.e.,carotid stenosis ≥ 50% associated with ipsilateral transient or visual TIA evidenced by amaurosis fugax, ipsilateral hemispheric TIAs or ipsilateral stroke within 6 months).

5. Prior occlusion of LAA.

6. The patient has an implanted mechanical mitral valve.

7. The patient requires long-term warfarin therapy due to:

1. Secondary to conditions such as prior arterial embolism or other indications such as pulmonary embolism or deep vein thrombosis within the previous 6 months
2. The patient is in a hypercoaguable state; exclude the patient if per medical record documentation, the patient meets any of the following criteria:

   * Thrombosis occurring ≤ 40 years of age
   * Idiopathic or recurrent VTE (venous thrombo-embolism)
   * Thrombosis at an unusual site (cerebral veins, hepatic veins, renal veins, IVC, mesenteric veins)
   * Family history of VTE or of inherited prothrombotic disorder, recurrence/extension of thrombosis while adequately anticoagulated.

     8. The patient is actively enrolled in another trial of a cardiovascular device or an investigational drug (post-market study participation and registries are acceptable).

     9. The patient is pregnant or pregnancy is planned during the course of the investigation if patient is of child bearing potential.

     10. Any clinically significant medical condition or presence of any laboratory abnormality prior to randomization that is considered by the investigator to be clinically important and could interfere with the conduct of the study or not meeting procedure guidelines for TAVR or WATCHMAN.

     11. The patient has a life expectancy of less than two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Kapadia, MD, Principal Investigator — The Cleveland Clinic
Locations (32):
- United States (32):
  - Banner University Medical Center, Phoenix, Arizona
  - Sutter Health/Palo Alto Medical Foundation, Burlingame, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - UCHealth Medical Center of the Rockies, Loveland, Colorado
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Baptist Health Jacksonville, Jacksonville, Florida
  - Northside Hospital, St. Petersburg, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Prairie Cardiovascular Consultants, Springfield, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - St. Vincent Heart Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension St. John Hospital, Detroit, Michigan
  - Medstar Washington University, St Louis, Missouri
  - CHI Health Research Center, Omaha, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - University at Buffalo, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - The Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Pinnacle Health, Wormleysburg, Pennsylvania
  - WellSpan York Hospital, York, Pennsylvania
  - Lexington Cardiology, West Columbia, South Carolina
  - Austin Heart, Austin, Texas
  - Heart Hospital Baylor Plano, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Aspirus Research Institute, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kapadia SR, Krishnaswamy A, Whisenant B, Potluri S, Iyer V, Aragon J, Gideon P, Strote J, Leonardi R, Agarwal H, Larrain G, Sanchez C, Panaich SS, Harvey J, Vahl T, Menon V, Wolski K, Wang Q, Leon MB. Concomitant Left Atrial Appendage Occlusion and Transcatheter Aortic Valve Replacement Among Patients With Atrial Fibrillation. Circulation. 2024 Mar 5;149(10):734-743. doi: 10.1161/CIRCULATIONAHA.123.067312. Epub 2023 Oct 24. PMID 37874908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: General study population consisted of patients having non-valvular Atrial Fibrillation undergoing standard of care TAVR. Recruitment started December 2017 with the final subject enrolled November 2020. Only medical centers with approval for commercial WATCHMAN implantation were included in this trial. There were 34 North American sites in the WATCH TAVR trial.
Groups:
- TAVR + Medical Therapy: n=175 will undergo Transcatheter Aortic Valve Replacement (TAVR) alone with medical management for atrial fibrillation
  TAVR: Transcatheter Aortic Valve Replacement
- TAVR + WATCHMAN: n=175 will undergo simultaneous Transcatheter Aortic Valve Replacement (TAVR) with a WATCHMAN device.
  WATCHMAN: WATCHMAN Device is composed of a self-expanding nitinol structure with a porous membrane on the proximal face. The implant device is delivered to the Left Atrial Appendage by femoral venous access and transseptal puncture to enter the left atrium.
  TAVR: Transcatheter Aortic Valve Replacement
Period: Overall Study
Arm/Group | TAVR + Medical Therapy | TAVR + WATCHMAN
Started (Enrollment started December 2017. Last subject enrolled November 2020. Subjects were followed for 24 months from enrollment date. Follow up period ended December 2022.) | 172 | 177
Completed | 172 | 177
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants in number
Groups:
- Total: Total of all reporting groups
Arm/Group | TAVR + Medical Therapy | TAVR + WATCHMAN | Total
Number analyzed (Participants) | 172 | 177 | 349
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 172 | 177 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.5 (6.4) | 80.8 (7.8) | 81.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 69 | 135
  Male | 106 | 108 | 214
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 167 | 173 | 340
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 172 | 177 | 349

OUTCOME MEASURES:

1. Primary Outcome: Composite of All-cause Mortality, Stroke and Bleeding
Description: First occurrence of all-cause mortality, stroke (ischemic or hemorrhagic), or bleeding (life-threatening and major) events through 2 years post-randomization.
Time Frame: Through 2 year post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | TAVR + Medical Therapy | TAVR + WATCHMAN
Number analyzed (Participants) | 172 | 177
Participants | 60 | 64

2. Secondary Outcome: All-cause Mortality
Description: All deaths through 2 year
Time Frame: Through 2 year post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | TAVR + Medical Therapy | TAVR + WATCHMAN
Number analyzed (Participants) | 172 | 177
Participants | 39 | 37

3. Secondary Outcome: Stroke
Description: First occurrence of any ischemic or hemorrhagic stroke through 2 year
Time Frame: Through 2 year post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | TAVR + Medical Therapy | TAVR + WATCHMAN
Number analyzed (Participants) | 172 | 177
Participants | 12 | 10

4. Secondary Outcome: Bleeding
Description: First occurrence of any life-threatening or major bleeding through 2 year
Time Frame: Through 2 year post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | TAVR + Medical Therapy | TAVR + WATCHMAN
Number analyzed (Participants) | 172 | 177
Participants | 30 | 35

5. Other Pre Specified Outcome: Cardiovascular Mortality
Description: Cardiovascular related mortality through 2 year
Time Frame: Through 2 year post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | TAVR + Medical Therapy | TAVR + WATCHMAN
Number analyzed (Participants) | 172 | 177
Participants | 22 | 20

6. Other Pre Specified Outcome: Thrombus or Embolism
Description: Incidence of arterial or venous embolism
Time Frame: Through 2 year post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | TAVR + Medical Therapy | TAVR + WATCHMAN
Number analyzed (Participants) | 172 | 177
Participants | 3 | 16

7. Other Pre Specified Outcome: Re-hospitalization
Description: Incidence of re-hospitalizations related to the WATCHMAN procedure or WATCHMAN device
Time Frame: Through 2 year post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | TAVR + Medical Therapy | TAVR + WATCHMAN
Number analyzed (Participants) | 172 | 177
Participants | 22 | 18

8. Other Pre Specified Outcome: Quality of Life Score: KCCQ-12
Description: Change from baseline in quality of life (QoL) as measured using the KCCQ-12 score. Kansas City Cardiomyopathy Questionnaire (KCCQ-12) is a validated tool used to assess heart failure and how it affects the participant's life. Four domain scores and one summary score are generated from the KCCQ-12: Physical Limitation Score, Symptom Frequency Score, Quality of Life Score, Social Limitation Score and a Summary Score. Scale ranges for each question 1 to 6 (Extremely limited 1, Quite a bit limited 2, Moderately limited 3, Slightly limited 4, Not at all limited 5, Limited for other reasons or did not do the activity 6. The Summary score represents an integration of the patient's physical limitation, symptom frequency, quality of life and social limitation. The total score is calculated as the average of the above scale descriptions. Scores are scaled 0-100, where 0 denotes the lowest reportable health status. Scores of 100 indicate the highest reportable health better outcome status.
Time Frame: Through 2 year post-randomization
Population: Patient's with non missing KCCQ data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAVR + Medical Therapy | TAVR + WATCHMAN
Number analyzed (Participants) | 169 | 176
score on a scale
  KCCQ Questionnaire Score Visit 1-Baseline | 39.77 (15.55) | 40.8 (15.21)
  KCCQ Questionnaire Score Visit 2- 45 Days: number analyzed (Participants) | 165 | 171
  KCCQ Questionnaire Score Visit 2- 45 Days | 55.2 (17.77) | 55.1 (17.94)
  KCCQ Questionnaire Score (Visit 3- 6 Months): number analyzed (Participants) | 147 | 164
  KCCQ Questionnaire Score (Visit 3- 6 Months) | 56.6 (17.97) | 57.61 (15.18)
  KCCQ Questionnaire Score (Visit 4-12 Months): number analyzed (Participants) | 118 | 147
  KCCQ Questionnaire Score (Visit 4-12 Months) | 56.3 (18.42) | 57.4 (15.67)
  KCCQ Questionnaire Score (Visit 5- 24 months): number analyzed (Participants) | 120 | 137
  KCCQ Questionnaire Score (Visit 5- 24 months) | 57.1 (18.99) | 57.0 (16.51)

9. Other Pre Specified Outcome: Procedural Costs
Description: Procedural costs related to the initial TAVR and WATCHMAN procedures
Time Frame: Mean cost during hospitalization up to 40 days.
Population: Sites willing to provide cost data.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | TAVR + Medical Therapy | TAVR + WATCHMAN
Number analyzed (Participants) | 25 | 21
dollars | 195309.64 (206704.690) | 216020.41 (91603.542)

ADVERSE EVENTS:
Time Frame: Events collected within two years following randomization.
Arm/Group | TAVR + Medical Therapy | TAVR + WATCHMAN
All-Cause Mortality (participants affected / at risk) | 39/172 | 37/177
Serious Adverse Events (participants affected / at risk) | 90/172 | 87/177
Other Adverse Events (participants affected / at risk) | 131/172 | 127/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAVR + Medical Therapy (N=172) | TAVR + WATCHMAN (N=177)
Cardiac - Other (Cardiac disorders) | 26 | 29
Bleeding - Event Associated with bleeding (Blood and lymphatic system disorders) | 26 | 31 — Event associated with bleeding
Cardiac - Heart Failure (Cardiac disorders) | 7 | 18 — Heart Failure
Renal - Other (not bleeding) (Renal and urinary disorders) | 6 | 8 — Other- not bleeding
Infection - Other (except endocarditis and device infection) (Infections and infestations) | 7 | 9 — Other (except endocarditis and device infection)
Cardiac - Sudden Cardiac Death/Cardiac Arrest (Cardiac disorders) | 8 | 5 — Sudden Cardiac Death/Cardiac Arrest
Any AE with symptoms that could possibly be contributed to WATCHMAN or TAVR device/procedure (General disorders) | 4 | 9
Anemia (Blood and lymphatic system disorders) | 6 | 4 — Not associated with bleeding
Cancer/Malignancy (General disorders) | 4 | 6
Pulmonary - Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Neurologic - Ischemic Stroke (Nervous system disorders) | 3 | 5
Pulmonary - Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 — Pleural Effusion (not sanguineous)
Neurologic - Other (Nervous system disorders) | 4 | 3 — Other
Neurologic - Stroke Type Unknown (Nervous system disorders) | 5 | 1 — Stroke Type Unknown
Trauma (General disorders) | 1 | 4
Renal - AKI (requiring dialysis) (Renal and urinary disorders) | 4 | 2
Cardiac - Pericardial Effusion (not hemorrhagic) (Cardiac disorders) | 3 | 2 — Pericardial Effusion (not hemorrhagic)
COVID-19 Infection (Infections and infestations) | 2 | 3
Rehospitalization related to TAVR device or procedure (General disorders) | 3 | 2
Infection - UTI (Infections and infestations) | 2 | 2 — UTI
Thrombosis - Other systemic (Vascular disorders) | 1 | 3 — Other systemic (other than stroke)
GI- Other (not bleeding) (Gastrointestinal disorders) | 0 | 3 — Other (not bleeding)
Cardiac - Endocarditis (Cardiac disorders) | 2 | 2
COD Unknown (General disorders) | 4 | 0
Pulmonary - Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 — Embolism
Neurologic - TIA (Nervous system disorders) | 2 | 1 — TIA
Cardiac - Myocardial Infarction (Cardiac disorders) | 3 | 0
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 1 — Other
Cardiac - AV Regurgitation/Leak (Cardiac disorders) | 2 | 0 — AV Regurgitation/Leak
Thrombosis - WATCHMAN Device (Vascular disorders) | 0 | 2 — WATCHMAN Device
Thrombus- Atrial (not arterial) (Cardiac disorders) | 0 | 2 — Atrial (not arterial)
Septic Shock (General disorders) | 1 | 1
Endocrine Disorders (Endocrine disorders) | 1 | 1
Cardiac - Angina/Chest Pain/CAD (Cardiac disorders) | 1 | 1
Pulmonary - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — Pneumonia
Pulmonary - COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — COPD
Neurologic - Subdural Hematoma (Nervous system disorders) | 1 | 0
Vascular Pseudoaneurysm (Vascular disorders) | 1 | 0 — Requires endovascular repair
Vascular AV Fistula (intervention required) (Vascular disorders) | 1 | 0
Neruo- Mental Status Changes/Confusion (not stroke or TIA) (Nervous system disorders) | 0 | 1 — Mental Status Changes/Confusion (not stroke or TIA)
Cardiac - Heart Valve Damage (Cardiac disorders) | 1 | 0
Thrombosis - Venous (including DVT) (Vascular disorders) | 0 | 1 — Venous (including DVT)
Thrombosis - TAVR Device (Vascular disorders) | 0 | 1 — TAVR Device
Thrombosis - Other NON Cardiac Device (Vascular disorders) | 0 | 1 — Other NON Cardiac Device
Hypokalemia (General disorders) | 1 | 0
Supra-therapeutic INR (General disorders) | 0 | 1
Hepatobiliary (not bleeding) (General disorders) | 0 | 1
Rehospitalization related to WATCHMAN procedure or device (not listed above) (General disorders) | 0 | 1
Device Embolization - Catheter Retrieval (General disorders) | 0 | 1
Cardiac - Heart Valve Damage (Cardiac disorders) | 1 | 0 — Heart Valve Damage
Thrombosis- Venous (including DVT) (Vascular disorders) | 0 | 1 — Venous (including DVT)
Thrombosis - TAVR Device (Vascular disorders) | 0 | 1
Rehospitalization related to WATCHMAN procedure or device (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAVR + Medical Therapy (N=172) | TAVR + WATCHMAN (N=177)
Bleeding (Blood and lymphatic system disorders) | 54 | 57 — Event Associated with bleeding
Cardiac - Other (Cardiac disorders) | 40 | 57 — Cardiac- Other
Rental (Renal and urinary disorders) | 6 | 8 — Other- not bleeding
Trauma (General disorders) | 10 | 10
Infection (Infections and infestations) | 11 | 14 — Other (except endocarditis and device infection)
Anemia (Blood and lymphatic system disorders) | 12 | 7 — Not associated with bleeding
Any AE with symptoms that could possibly be contributed to WATCHMAN or TAVR device/procedure (General disorders) | 8 | 12 — Any AE with symptoms that could possibly be contributed to WATCHMAN or TAVR device/procedure
Neurologic (Nervous system disorders) | 8 | 10 — Other
Infection - UTI (Renal and urinary disorders) | 6 | 5 — UTI
Cancer/Malignancy (General disorders) | 5 | 9
Cardiac - Sudden Cardiac Death/Cardiac Arrest (Cardiac disorders) | 9 | 5 — Cardiac - Sudden Cardiac Death/Cardiac Arrest
Neurologic - Ischemic Stroke (Nervous system disorders) | 6 | 8 — Ischemic Stroke
Neurologic - TIA (Nervous system disorders) | 7 | 4 — TIA
Pulmonary - Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Cardiac - Angina/Chest Pain/CAD (Cardiac disorders) | 5 | 5 — Angina/Chest Pain/CAD
Pulmonary - Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 1 — Pleural Effusion (not sanguineous)
COVID-19 Infection (Infections and infestations) | 4 | 4
Pulmonary - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 | 2
COD Unknown (General disorders) | 6 | 2
Cardiac - Pericardial Effusion (not hemorrhagic) (Cardiac disorders) | 4 | 3 — Pericardial effusion (not hemorrhagic)
Neurologic - Stroke Type Unknown (Nervous system disorders) | 6 | 1 — Stroke Type Unknown
Neurologic - Mental Status Changes/Confusion (Nervous system disorders) | 3 | 4 — Mental Status Changes/Confusion (not stroke or TIA)
Thrombosis - Venous (including DVT) (Vascular disorders) | 3 | 3 — Venous (including DVT)
Renal- AKI (requiring dialysis) (Renal and urinary disorders) | 4 | 2 — AKI (requiring dialysis)
Rehospitalization related to TAVR device or procedure (not listed) (General disorders) | 4 | 2 — Related to TAVR device or procedure (not listed)
Thrombus - Atrial (not arterial) (Vascular disorders) | 0 | 6
Cardiac - Endocarditis (Cardiac disorders) | 2 | 2
GI- Other (not bleeding) (Gastrointestinal disorders) | 0 | 4
Cardiac - Myocardial Infarction (Cardiac disorders) | 3 | 1 — Myocardial infarction
Thrombosis - Other Systemic (other than stroke) (Vascular disorders) | 1 | 3
Hypokalemia (Blood and lymphatic system disorders) | 2 | 2
Endocrine Disorders (Endocrine disorders) | 2 | 1
Pulmonary - Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Neurologic - Subdural Hematoma (Nervous system disorders) | 2 | 0
Cardiac - AV Regurg/Leak (Cardiac disorders) | 2 | 0
Vascular Pseudoaneurysm (Vascular disorders) | 2 | 0 — no intervention required
Thrombosis - WATCHMAN Device (Vascular disorders) | 0 | 2
Septic Shock (Infections and infestations) | 1 | 1
Cardiac - Atrial Septal Defect (latrogenic) (Cardiac disorders) | 0 | 2 — Atrial Septal Defect (latrogenic)
Device Embolization - Catheter Retrieval (Vascular disorders) | 0 | 2 — Catheter Retrieval
Pulmonary - COPD (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Vascular Pseudoaneurysm (Vascular disorders) | 1 | 0 — requires endovascular repair
Vascular AV Fistual (Vascular disorders) | 1 | 0 — intervention required
Neoplasm Benign & Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Incl Cysts and Polyps
Leukocytosis (General disorders) | 0 | 1
Cardiac - Heart Valve Damage (Cardiac disorders) | 1 | 0 — Heart Valve Damage
Inflammatory/Immunologic (Infections and infestations) | 1 | 0
Thrombosis - TAVR Device (Vascular disorders) | 0 | 1
Vascular AV Fistula (Vascular disorders) | 0 | 1 — no intervention required
Thrombosis - Other NON Cardiac Device (Vascular disorders) | 0 | 1 — Other NON Cardiac Device
Thrombosis - Other Cardiac Device (Vascular disorders) | 0 | 1
Supra-therapeutic INR (General disorders) | 0 | 1
Hepatobiliary (not bleeding) (Hepatobiliary disorders) | 0 | 1 — not bleeding
Rehospitalization related to WATCHMAN procedure or device (General disorders) | 0 | 1 — Related to WATCHMAN procedure or device
Pancreatic (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT03173534/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT03173534/SAP_001.pdf
  • Informed Consent Form (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT03173534/ICF_002.pdf